CLINICAL TRIAL: NCT04459013
Title: Evaluation of the Release of Monomers From Composite Bonding Resins in Orthodontics
Acronym: MONORTHO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200328
Record Dates: First submitted 2020-06-17; First posted 2020-07-07 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Dent Disease
Keywords: Bisphenol A; toxicity; Composite; orthodontic retainers; release; endocrine disruptors
MeSH Terms: conditions — Dent Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient of the orthodontic consultation
  Interventions: Other: Salivary samples

INTERVENTIONS:
Other: Salivary samples — The salivary samples will be collected at 5 defined times

SUMMARY:
In recent decades, the field of public health has become increasingly interested in endocrine disruptors, and their effects on humans. Indeed, various scientific studies have highlighted an evolution in the frequency of pathologies due to these substances, affecting in particular the reproductive organs. Many concerns are expressed about the impact of these substances, present in the environment or in consumer products, on the hormonal system. Effects have been observed in animals in experimental studies, but the question of extrapolating these results to humans arises, especially for exposures at low doses.

In orthodontics, the composite is the material of choice mainly for bonding fasteners, then bonding a compression wire. These composite materials contain many monomers. The polemics launched on Bisphenol A and the questions of our patients on the nature and toxicity of dental products oblige us to reflect on their harmfulness after their placement in the oral cavity. Many questions arise today about dental composites and their participation in the release of endocrine disruptors. Indeed, Bisphenol A is used in the manufacturing process of the monomers of orthodontic composites, as precursors of Bis-GMA and Bis-DMA. The objective of this study is to search for the presence of BPA, TEGDMA, BisGMA, BisDMA and UDMA monomers, and to carry out the samples and their analysis at different clinical times (at T0, after the removal of orthodontic attachments, after the placement of the compression, one hour later, one week later, one month later and 6 months later) and the comparison of this quantification to that without orthodontic restraint. Studies have been performed in vitro, but very little in vivo. In addition, these studies are only carried out on release at the time of installation, but few are interested in the continuation of the phenomenon over time and the deterioration of the composite. Although the short-term toxicity of BPA is low, its dangerousness lies in its potential endocrine disrupting effect and which can induce long-term chronic toxicity.

Compounds such as TEGDMA, BisGMA, BisDMA and UDMA differ greatly in their volatility due to their different chemical structures as well as in their stability in saliva; Many methods have been developed to study each monomer individually or to study them simultaneously using different analytical techniques to determine their presence and to quantify them after their release from dental products. The analysis of the samples is carried out by liquid chromatography (HPLC).

DETAILED DESCRIPTION:
For several years, we have been wondering about the potential deleterious effects of bisphenol A (BPA) on our organism. Known as an endocrine disruptor, its action has been demonstrated at different levels of the human body and by different mechanisms. Its endocrine activity is due to its structure close to that of estradiol. Cytotoxicity is the property of a chemical or biological agent to be toxic to cells, possibly destroying it. Bisphenol A (BPA) has received increasing attention in recent years. It is used in the monomer manufacturing process of composites customary in orthodontics, as a precursor of Bis-DMA and Bis-GMA, but is not normally found in pure form in these composites. In the mouth, these materials are subject to numerous degradation constraints, initial and long-term: thermal variations, pH change, mechanical wear, enzymatic, bacterial and salivary attack. They are therefore responsible for the possible release of BPA, found in many human biological fluids, including saliva. The monomers present in the composite resins are released in 2 stages: immediate release where the non-polymerized monomers are found in the saliva for a few hours after the treatment, delayed release where the monomers can be released following the treatment by the various mechanisms of wear and degradation of the composite. If the BPA is mainly released in saliva within three hours after the establishment of the dental restoration, the long-term release remains to be determined, which explains the patient's follow-up time of 6 months.

The main objective of this research is the quantification of the Bisphenol A monomer released during the placement of a mandibular orthodontic compression in order to raise awareness among professionals and the comparison of this quantification to that without orthodontic restraint. The study relates to the analysis of patients followed in the dental department at the Pitié Salpetrière hospital. The study briefing note will be presented to patients during the visit. Non-opposition will be collected and notified in the patient's medical file after a 15-day cooling-off period.

The salivary samples will be collected at 5 defined times: before removal of the orthodontic brackets (T0), after removal (T1), just after application of the compression (T2), then at one hour (T3), one month (T4) and 6 months (T5), as part of the end of their orthodontic treatment. Control samples will be taken from patients who do not have a composite restoration in their mouth. The inclusion criteria are patients undergoing orthodontic treatment (multi-attachment device) with planned debagging and requiring compression with mandibular bonded wire from canine to canine and maxillary groove, without composite restoration in the mouth, with good hygiene and not gingival inflammation. The exclusion criteria are patients requiring maxillary bonded compression, with composite restoration in the mouth, carious lesions, smokers, with chronic pathologies and / or drugs, with chronic exposure to Bisphenol A (construction sites, service stations ... ). The composite cartridges will be weighed before and after their use, to have the exact quantity of material placed in the mouth. For laying the compression wire, the protocol will also be identical to the bonding protocol in adhesive dentistry.

The samples are analyzed by liquid chromatography (HPLC) on the Bioprofiler platform (Metabolism Platform) of the Functional and Adaptive Biology Unit - CNRS UMR 8251 at Paris Diderot University.

The analytical method chosen for the identification and quantification of the compounds is high pressure liquid chromatography (HPLC). This method allows the separation of the constituents of a very complex mixture. The HPLC consists of two pumps which maintain a mobile phase under pressure in a column (stationary phase). The sample is injected into the circulation system of the mobile phase and passes into the column where the different constituents are more or less retained. The nature of the mobile phase and of the column allows separation according to the physicochemical properties of the constituents of a mixture.

Developments and optimizations of extraction and dosage methods allowing the analysis of the release of bisphenols by orthodontic materials in saliva samples were carried out on this platform.

ELIGIBILITY:
Inclusion Criteria common to both groups:

* Patient of the orthodontic consultation consultant in the dentistry department of the Pitié Salpêtrière hospital,
* Information and collection of the non-opposition of the adult patient or representatives of the parental authority for minors
* Good dental hygiene at the discretion of the investigator
* Patient agreeing to be followed for 6 months
* Good written and oral comprehension of the French language

case-specific:

* Age between 10 and 70 years inclusive,
* Patients undergoing orthodontic treatment (multi-attachment device) with planned debagging and requiring compression with bonded mandibular wire from canine to canine, and maxillary groove

Specific to witnesses:

* Age between 18 and 70 inclusive
* Patients undergoing orthodontic treatment (multi-attachment appliance) with planned debridement without the need for a retainer

Exclusion Criteria common to both groups:

* Under tutorship or curatorship
* Opposition of the minor patient
* Gingival inflammation
* Patients requiring maxillary bonded restraint
* Composite restoration in the mouth
* Carious lesions
* Smokers
* Patients with chronic pathologies and / or under medication
* Chronic exposure to Bisphenol A.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient of the orthodontic consultation consultant in the dentistry department of the Pitié Salpêtrière hospital,
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Changement of quantity of the Bisphenol A | before any medical procedure, and regularly after the medical procedure
  The main objective of this research is the quantification of the Bisphenol A monomer released during the placement of a mandibular orthodontic compression in order to raise awareness among professionals or without orthodontic restraint..

SECONDARY OUTCOMES:
Changement of quantity of the release of TEGDMA monomers; UDMA; BisGMA and BisDMA | before any medical procedure, and regularly after the medical procedure
  The secondary objective of this study is the quantification of the release of TEGDMA monomers; UDMA; BisGMA and BisDMA by orthodontic materials in saliva samples.
Changement of those quantities in patients with mandibular orthodontic restraints with patients without restraints | before any medical procedure, and regularly after the medical procedure
  - High pressure liquid chromatography (HPLC) quantification in "controls" of bisphenol A monomer released in saliva samples, TEGDMA, UDMA, BisGMA and BisDMA monomers

CONTACTS AND LOCATIONS:
Locations (1):
- Service Odontology, Hôpital Pitié-Salpêtrière, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No